CLINICAL TRIAL: NCT03490630
Title: Patient Reported Outcome After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09d (bariatric ss)
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Analgesia; Bariatric Surgery
Keywords: patient reported outcome; postoperative pain; pain related impairment; quality of life; prospective association study
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood (plasma and cells) or mucosal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients undergoing elective surgery with anesthesia

SUMMARY:
Prospective association study to analyse patients' outcome after bariatric surgery.

Outcome comprises postoperative pain, analgesia, postoperative side-effects, long-lasting pain, patients' impairment in daily living.

DETAILED DESCRIPTION:
Background

Bariatric surgery is a common procedure. Data on patient related outcome beyond loss of body weight are scarce. The question arises which patient is at specific risk for an unfavorable outcome after bariatric surgery.

Objective

The aim of this study is to investigate variables possibly associated with impaired outcome and increased patients' interference after bariatric surgery. Which patients are at risk for clinically meaningful impaired daily living?

Methods

Patients will be enrolled in a prospective observational study. Data will be collected in a registry with documentation of patient, surgery, anesthesia and analgesia related variables including preoperative status and postoperative patient reported outcome with a follow-up period up to 5 years after bariatric surgery.

Patients fill in standardized validated outcome questionnaires at predefined time points. The registry provides the basis for large scale analyses and benchmarks for several parameters.

Variables to be considered are pain scores after surgery, patient reported outcome, pain related interference after surgery (Brief Pain Inventory), quality of life (SF-12), long-term outcome, chronic (neuropathic) postsurgical pain, BMI, psychological questionnaires, surgery and patient related variables, including genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Elective bariatric surgery
* Patients' ability to understand the purpose of the study

Exclusion Criteria

* No informed consent
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2011-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
What influences pain related impairment after bariatric surgery | First day after surgery
  Measured by the validated International Pain Outcomes Questionnaire: Patient reported outcome using the numeric rating scale 0-10 (0=no impairment, 10=worst experience possible). Patients with severe pan (pain scores of NRS 6 and higher) are compared to those with no and mild pain.

SECONDARY OUTCOMES:
Change in pain related outcome after bariatric surgery | Up to 12 months after surgery
  Measurement of patient reported outcome by the BPI (Brief Pain Inventory). The BPI gives information on the physical and affective interference as well as pain scores using the numeric rating scale (NRS: 0-10). Cut-offs discussed for the three groups no/mild interference, moderate interference and severe interference are mean NRS-scores of 3 and 5.
Change in interference with daily activities after bariatric surgery | Up to to 5 years after surgery
  Physical and affective interference as well as pain scores measured by the Brief Pain Inventory (BPI). Independent variables e.g. Hospital Anxiety and Depression Scale (HADS) and further validated psychological questionnaires
Change in quality of life after bariatric surgery | Up to 5 years after surgery
  Measured by the 12 item short-form health survey (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike M Stamer, Prof. MD, Principal Investigator — Department of Anaestheisology and Pain Medicine, Inselspital, University of Bern; Frank Stüber, Study Director — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland